CLINICAL TRIAL: NCT00898157
Title: Analysis of E4494 Tissues to Determine the Prognostic Significance of Biomarkers in Diffuse Large B Cell Lymphoma (DLBCL) Treated With Standard Chemotherapy (CHOP) Plus Rituximab ®)1
Brief Title: Study of Biomarkers Using Tissue Samples From Older Patients With Diffuse Large B-Cell Lymphoma Treated With Combination Chemotherapy With or Without Rituximab on Clinical Trial ECOG-E4494
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000571530; ECOG-E4494T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Lymphoma
Keywords: contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; recurrent adult diffuse large cell lymphoma; stage I adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. It may also help doctors understand how patients respond to treatment.

PURPOSE: This laboratory study is looking at biomarkers using tissue samples from older patients with diffuse large B-cell lymphoma treated with combination chemotherapy with or without rituximab on clinical trial ECOG-E4494.

DETAILED DESCRIPTION:
OBJECTIVES:

* To construct tissue microarrays (TMA) using tissue samples from older patients with diffuse large B-cell lymphoma treated with standard CHOP chemotherapy (cyclophosphamide, doxorubicin, vincristine, and prednisone) with or without rituximab on clinical trial ECOG-E4494.
* To allow this TMA resource to be included in a large international effort (the Lunenburg Lymphoma Biomarker Consortium [LLBC]), partnering with several other similar randomized trials (EORTC, HOVON, GELA, MINT) in order to properly power and bring standardization to the study of biomarkers in lymphoma.
* To evaluate the clinical impact and prognostic importance of a number of biomarkers, including Bcl-2, Bcl-6, CD10, FOXP1, MUM1, Ki-67, CD5, and HLA-Dr.
* To determine the prognostic impact of clinical International Prognostic Index (IPI) variables in a large international study.
* To determine the relationship between different biomarkers and clinical predictors.
* To establish the TMA (using tissue samples from patients treated on clinical trial ECOG-E4494) as a resource for future ECOG-driven studies and for validation of novel biomarkers as they become recognized and available.

OUTLINE: Patients are stratified according to prior treatment (CHOP chemotherapy [cyclophosphamide, doxorubicin, vincristine, and prednisone] or CHOP-like chemotherapy vs CHOP chemotherapy with or without rituximab).

Tissue microarrays will be constructed using tissue samples previously collected from patients treated on clinical trial ECOG-E4494. Tissue microarrays will be used for biomarker studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of diffuse large B-cell lymphoma
* Received treatment on clinical trial ECOG-E4494

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients participating in E4494
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Actual)
Dates: Start 2007-09-24 (Actual); Primary Completion 2008-09-24 (Actual); Study Completion 2008-09-24 (Actual)

PRIMARY OUTCOMES:
Correlation of biomarkers with response and outcome | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Randall D. Gascoyne, MD, Study Chair — British Columbia Cancer Agency

REFERENCES:
- [Background] Habermann TM, Weller EA, Morrison VA, Gascoyne RD, Cassileth PA, Cohn JB, Dakhil SR, Woda B, Fisher RI, Peterson BA, Horning SJ. Rituximab-CHOP versus CHOP alone or with maintenance rituximab in older patients with diffuse large B-cell lymphoma. J Clin Oncol. 2006 Jul 1;24(19):3121-7. doi: 10.1200/JCO.2005.05.1003. Epub 2006 Jun 5. PMID 16754935
- [Result] Aurora V, Li S, Horning SJ, et al.: Prognostic significance of p53/p21 expression in DLBCL treated with CHOP or R-CHOP: a correlative study of E4494. [Abstract] J Clin Oncol 25 (Suppl 18): A-8038, 450s, 2007.
- [Result] Winter JN, Weller EA, Horning SJ, Krajewska M, Variakojis D, Habermann TM, Fisher RI, Kurtin PJ, Macon WR, Chhanabhai M, Felgar RE, Hsi ED, Medeiros LJ, Weick JK, Reed JC, Gascoyne RD. Prognostic significance of Bcl-6 protein expression in DLBCL treated with CHOP or R-CHOP: a prospective correlative study. Blood. 2006 Jun 1;107(11):4207-13. doi: 10.1182/blood-2005-10-4222. Epub 2006 Jan 31. PMID 16449523